CLINICAL TRIAL: NCT00003135
Title: A Phase I-II Trial of Mild Whole-Body Hyperthermia Combined With Liposomal Doxorubicin/5-Fluorouracil in Patients With Advanced Malignancy
Brief Title: Whole Body Hyperthermia Combined With Chemotherapy in Treating Patients With Metastatic Breast, Ovarian, Endometrial, or Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Joan M.C. Bull, University of Texas Health Science Center at Houston
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065903; UTHSC-MS-96205; NCI-V97-1356
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2009-04-30 (Estimated); Status verified 2008-12

CONDITIONS: Breast Cancer; Cervical Cancer; Endometrial Cancer; Ovarian Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; recurrent cervical cancer; stage IVB cervical cancer; stage IVA cervical cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; stage IV endometrial carcinoma; recurrent endometrial carcinoma; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Breast Neoplasms, Male | interventions — Fluorouracil; Diathermy

INTERVENTIONS:
Drug: fluorouracil
Drug: pegylated liposomal doxorubicin hydrochloride
Procedure: hyperthermia treatment

SUMMARY:
RATIONALE: Hyperthermia therapy kills tumor cells by heating them to several degrees above body temperature. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with hyperthermia may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving fluorouracil and liposomal doxorubicin together with systemic hyperthermia works in treating patients with metastatic breast, ovarian, endometrial, or cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate tumor response and toxicity induced by fluorouracil and doxorubicin HCl liposome combined with mild systemic hyperthermia in patients with metastatic breast, ovarian, endometrial, or cervical cancer.

OUTLINE: This is a time-escalation study of systemic hyperthermia.

Patients receive fluorouracil IV continuously over 24 hours on days 1-5 and doxorubicin HCl liposome IV over 30 minutes on day 6. Beginning on day 7, patients receive heat applied for 6-24 hours (in 6-hour sequential treatments) using a mild hyperthermia-induction device. Treatment repeats every 4-5 weeks for a total of 4 courses. Patients who achieve less than a complete response but have no disease progression may receive additional courses of chemotherapy alone.

Cohorts of 5 patients receive escalating durations of hyperthermia until the recommended phase II duration is determined. The recommended phase II duration of hyperthermia is defined as the level preceding that at which 1 of 5 patients experiences measurable toxicity. (Phase I closed as of 9/28/01)

Patients are followed at 4 weeks and then every 6 months for 1 year.

PROJECTED ACCRUAL: A maximum of 34 patients will be accrued for this study within 48 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic breast, ovarian, endometrial, or cervical carcinoma
* Measurable and evaluable disease
* No brain metastases
* No hepatic involvement greater than 80%
* No lung involvement greater than 30%
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Not specified

Menopausal status:

* Not specified

Performance status:

* Zubrod 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute granulocyte count greater than 1,500/mm^3
* Platelet count greater than 90,000/mm^3
* Normal bone marrow cellularity on bone marrow biopsy
* Thrombin time less than 17 sec
* Fibrinogen greater than 200 mg/dL
* FSP less than 40
* No coagulopathy

Hepatic:

* Bilirubin less than 2.0 mg/dL
* SGPT less than 2 times normal
* PT less than 14 sec
* PTT less than 35 sec

Renal:

* BUN less than 25 mg/dL
* Creatinine clearance at least 45 mL/min

Cardiovascular:

* Normal cardiovascular system
* Resting ventricular ejection fraction greater than 40%
* No prior myocardial infarction
* No symptomatic coronary artery disease
* No unstable blood pressure
* No thromboembolic disease

Neurologic:

* No seizures or other CNS disorders
* Negative computerized tomographic scan of brain

Pulmonary:

* FEV_1 greater than 70% of predicted
* Arterial pressure of oxygen greater than 60 mmHg on room air with appropriate pressure of carbon dioxide and pH values
* No history of cardiopulmonary or respiratory disease

Other:

* No other serious concurrent medical illness
* No diabetes mellitus

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior chemotherapy allowed

Endocrine therapy:

* No adrenal corticosteroids

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent cardiac glycosides, antianginal therapy, or antiarrhythmics
* No concurrent vasodilators, anticoagulants, thrombolytic agents, or aspirin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 1997-11; Primary Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Tumor response
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Joan M.C. Bull, MD, Study Chair — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States